CLINICAL TRIAL: NCT04867226
Title: Effectiveness of Colchicine Among Patients With COVID-19 Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hawler Medical University (Other)
Responsible Party: Principal Investigator, Aryan Mohamadfatih Jalal, Doctor Rheumatollogy, Hawler Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Effectiveness of colchicine
Record Dates: First submitted 2021-04-25; First posted 2021-04-30 (Actual); Last update posted 2021-06-22 (Actual); Status verified 2021-06

CONDITIONS: Coronavirus Infection
Keywords: covid-19, colchicine; Erbil,Iraq
MeSH Terms: conditions — Coronavirus Infections; COVID-19 | interventions — Colchicine; Therapeutics

STUDY DESIGN:
Intervention Model Description: 100 Patients will participate for eligibility and enroll in the study, an open labell randomize control clinical trial will held among patients who will infect with COVID-19 in whom they met the inclusion criteria, either treat at home with healthcare advises and follow up or at centres of COVID-19 in ERBIL city ( Rozhawa emergency hospital, Erbil international private hospital) .
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- colchicine drug (Active Comparator): participant in this group will be given a colchicine tablet alone or add to their Current treatment, Colchicine 0.5 mg twice daily (reduced to 0.5 mg/day, in patients with low body weight or develop side effect like gastrointestinal symptoms ),For 14 days or until symptoms subsides.
  Interventions: Drug: Colchicine 0.5 MG
- usual care (Active Comparator): control group will receive usual care COVID-19 treatment according to Iraqi protocol guideline and will not receive colchicine.
  Interventions: Drug: usual care treatment

INTERVENTIONS:
Drug: Colchicine 0.5 MG — participant will be given a Colchicine regimen in a dose of 0.5mg twice daily for 14 days or until symptoms subsides,those with low body weight and develop side effect like diarrhea and vomiting dose will be reduced and supportive treatment will be given .
  Other Names: colcrys; colchicum
  Arms: colchicine drug
Drug: usual care treatment — control group will receive usual care COVID-19 treatment according to Iraqi protocol guideline and will not receive colchicine.
  Other Names: treatment
  Arms: usual care

SUMMARY:
In November 2019, there were a lot of cases of an acute respiratory illness (then named at February 11th as COVID_19) which first case was reported in Wuhan, China,The SARS COV-2 had been spread in a fast way to involve whole world, As it's obvious that Colchicine is a drug that is most commonly and widely used to treat and prevent acute attacks of Gout, other crystal induced arthropathy,colchicine has important role in inhibiting activation of NLRP3 inflammasome these lead to decrease cytokine production , aim of study To evaluate whether colchicine is effective in the treatment of COVID-19 cases. And to measure the effectiveness of colchicine in alleviating and controlling pulmonary and extra pulmonary complications of COVID-19

DETAILED DESCRIPTION:
this is an open label, randomize control clinical trial ,the participant will be randomly assign in to two groups ( Group A and Group B), colchicine (group A) will treat with colchicine tablet alone or add to their Current treatment,Colchicine 0.5 mg twice daily (reduce to 0.5 mg/day, in patients with low body weight or develop side effects like gastrointestinal symptoms ),For 14 days or until symptoms subsides, while the control group will treat according to usual treatment guideline in COVID-19.

ELIGIBILITY:
Inclusion Criteria:

1.patients diagnosed clinically or by RT-PCR in nasopharyngeal swab specimens and/ or lung involvement confirm by computed tomography scan compatible with COVID-19patients 2.Age between 18 year and 70 years, 3.body weight > 50 kg, 4.with written informed consent from patients or relatives.

-

Exclusion Criteria 1 sensitivity to any medications of regimens, 2.e GFR less than 30. 3.pregnancy. 4.malignancy . 5.Participating in another clinical study and refusing to participate in the study at a later date or later, and they are already taking colchicine for other diseases .

-

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-05-08 (Actual); Primary Completion 2021-06-18 (Actual); Study Completion 2021-06-18 (Actual)

PRIMARY OUTCOMES:
need for supplemental oxygen | 14 days following randomization
  number of patients need supplemental oxygen
length of hospital stay | 14 days following randomization
  number of patients who admit to hospital and duration of stay
need for invasive mechanical ventilation | 14 days following randomization
  number of patients need invasive mechanical ventilation
death rate | 14 days following randomization
  number of patients who die during randomization

SECONDARY OUTCOMES:
oxygen saturation measurement | 14 days following randomization
  Sp02 measurement by pulse oximetry
musculoskeletal symptoms | 14 days following randomization
  participants who have back pain and myalgia measure by patient analogue scale of pain
change in severity marker | 14 days following randomization
  CRP measurement
change in inflammatory marker | 14 days following randomization
  ferritin
change in severity marker | 14 days following randomization
  D.Dimer
change in marker | 14 days following randomization
  leukocyte
adverse effect | 14 days following randomization
  number of participants who develop adverse effect with treatment

CONTACTS AND LOCATIONS:
Overall Officials: Dashty Albustany, MBChB.FRCP, Study Director — assistant professor in medicine,consultant Rheumatologist; Aryan MF Jalal, Principal Investigator — M.B.CH.B, doctor Rheumatology
Locations (1):
- Hawler medical university ,Rozhawa emergency hospital, Erbil, Iraq

REFERENCES:
- [Background] Lu H, Stratton CW, Tang YW. Outbreak of pneumonia of unknown etiology in Wuhan, China: The mystery and the miracle. J Med Virol. 2020 Apr;92(4):401-402. doi: 10.1002/jmv.25678. Epub 2020 Feb 12. No abstract available. PMID 31950516
- [Background] Vardhana SA, Wolchok JD. The many faces of the anti-COVID immune response. J Exp Med. 2020 Jun 1;217(6):e20200678. doi: 10.1084/jem.20200678. PMID 32353870
- [Background] Mehta P, McAuley DF, Brown M, Sanchez E, Tattersall RS, Manson JJ; HLH Across Speciality Collaboration, UK. COVID-19: consider cytokine storm syndromes and immunosuppression. Lancet. 2020 Mar 28;395(10229):1033-1034. doi: 10.1016/S0140-6736(20)30628-0. Epub 2020 Mar 16. No abstract available. PMID 32192578
- [Background] Wu C, Chen X, Cai Y, Xia J, Zhou X, Xu S, Huang H, Zhang L, Zhou X, Du C, Zhang Y, Song J, Wang S, Chao Y, Yang Z, Xu J, Zhou X, Chen D, Xiong W, Xu L, Zhou F, Jiang J, Bai C, Zheng J, Song Y. Risk Factors Associated With Acute Respiratory Distress Syndrome and Death in Patients With Coronavirus Disease 2019 Pneumonia in Wuhan, China. JAMA Intern Med. 2020 Jul 1;180(7):934-943. doi: 10.1001/jamainternmed.2020.0994. PMID 32167524
- [Background] Banu N, Panikar SS, Leal LR, Leal AR. Protective role of ACE2 and its downregulation in SARS-CoV-2 infection leading to Macrophage Activation Syndrome: Therapeutic implications. Life Sci. 2020 Sep 1;256:117905. doi: 10.1016/j.lfs.2020.117905. Epub 2020 Jun 3. PMID 32504757
- [Background] Alhogbani T. Acute myocarditis associated with novel Middle east respiratory syndrome coronavirus. Ann Saudi Med. 2016 Jan-Feb;36(1):78-80. doi: 10.5144/0256-4947.2016.78. PMID 26922692
- [Background] Bangalore S, Sharma A, Slotwiner A, Yatskar L, Harari R, Shah B, Ibrahim H, Friedman GH, Thompson C, Alviar CL, Chadow HL, Fishman GI, Reynolds HR, Keller N, Hochman JS. ST-Segment Elevation in Patients with Covid-19 - A Case Series. N Engl J Med. 2020 Jun 18;382(25):2478-2480. doi: 10.1056/NEJMc2009020. Epub 2020 Apr 17. No abstract available. PMID 32302081
- [Background] Wang D, Hu B, Hu C, Zhu F, Liu X, Zhang J, Wang B, Xiang H, Cheng Z, Xiong Y, Zhao Y, Li Y, Wang X, Peng Z. Clinical Characteristics of 138 Hospitalized Patients With 2019 Novel Coronavirus-Infected Pneumonia in Wuhan, China. JAMA. 2020 Mar 17;323(11):1061-1069. doi: 10.1001/jama.2020.1585. PMID 32031570
- [Background] Crittenden DB, Lehmann RA, Schneck L, Keenan RT, Shah B, Greenberg JD, Cronstein BN, Sedlis SP, Pillinger MH. Colchicine use is associated with decreased prevalence of myocardial infarction in patients with gout. J Rheumatol. 2012 Jul;39(7):1458-64. doi: 10.3899/jrheum.111533. Epub 2012 Jun 1. PMID 22660810
- [Background] Slobodnick A, Shah B, Krasnokutsky S, Pillinger MH. Update on colchicine, 2017. Rheumatology (Oxford). 2018 Jan 1;57(suppl_1):i4-i11. doi: 10.1093/rheumatology/kex453. PMID 29272515
- [Derived] Mikolajewska A, Fischer AL, Piechotta V, Mueller A, Metzendorf MI, Becker M, Dorando E, Pacheco RL, Martimbianco ALC, Riera R, Skoetz N, Stegemann M. Colchicine for the treatment of COVID-19. Cochrane Database Syst Rev. 2021 Oct 18;10(10):CD015045. doi: 10.1002/14651858.CD015045. PMID 34658014